CLINICAL TRIAL: NCT06513494
Title: A Stepped-wedge, Cluster, and Randomized Trial to Evaluate Active Health Education Methods to Increase Human Papillomavirus Vaccine Coverage in Youth
Brief Title: Active Health Education to Increase HPV Vaccine Coverage in Youth: A Stepped-wedge, Cluster, and Randomized Trial
Acronym: EDUCAVAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EDUCAVAC trial
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Vaccine Refusal; Vaccine Hesitancy
Keywords: vaccination coverage; HPV vaccine; stepped-wedge design; students
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Stepped-wedge, Cluster, and Randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Students Education plus Teacher Training (Experimental): Clusters will perform active training for both teachers and students.
  Interventions: Behavioral: Active Students Education plus Teacher Training
- Active Students Education (Experimental): Clusters will perform active training for only students.
  Interventions: Behavioral: Active Students Education
- Basic Health Unit Active Orientation (Experimental): Clusters will receive a nurse-led orientation session on vaccination for students in schools.
  Interventions: Behavioral: Basic Health Unit Active Orientation
- Usual care (Other): No project interventions will be carried out.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Active Students Education plus Teacher Training — The teacher undergoes 30 hours of self-instructional training on vaccination through an online platform tailored for the relevant age group. Additionally, students receive active vaccinations and health education over two months
  Arms: Active Students Education plus Teacher Training
Behavioral: Active Students Education — Students receive active vaccinations and health education over two months.
  Arms: Active Students Education
Behavioral: Basic Health Unit Active Orientation — Nurses from basic health units will conduct an active orientation session at schools about vaccination for students.
  Arms: Basic Health Unit Active Orientation
Other: Usual care — No project interventions will be carried out.
  Arms: Usual care

SUMMARY:
This study aims to evaluate the impact of active health education methodologies on increasing adherence to the HPV vaccine among schoolchildren. The project will involve 196 schools across Brazil, encompassing a total of 5,000 students.

A stepped-wedge implementation design will be applied, with clusters being randomized every two months to one of four interventions.

Each intervention will be implemented in 48 schools.

DETAILED DESCRIPTION:
The adherence to the HPV vaccine among young people has declined recently, particularly in Brazil. While previous studies have shown that interventions such as text messaging can increase vaccination coverage, there is still a lack of robust data on the effectiveness of direct interventions in school populations using active health education methods. This study aims to evaluate the impact of active health education methodologies on increasing adherence to the HPV vaccine among schoolchildren.

The project will involve 80 schools across Brazil, including a total of 5,000 students. These schools will be randomized into clusters of five.

The study will apply a stepped-wedge implementation design, with clusters being randomized every two months to one of four interventions:

Education for students and teachers training + Basic Health Unit action in schools Education for students without teachers training + Basic Health Unit action in schools Only Basic Health Unit activities Usual control

ELIGIBILITY:
Criteria for students

Inclusion Criteria:

* Students of both sexes aged 9 to 14 years old.

Exclusion Criteria:

* Students with a complete HPV vaccination (two doses) received.

Criteria for Clusters

Inclusion Criteria:

* The school has enrolled students aged 9 to 14 years old.

Exclusion Criteria:

* Schools that do not have students aged between 9 and 14;
* Schools that provided only distance education

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of children and adolescents with at least one dose of HPV vaccination following the intervention | 12 months
  Rate of HPV vaccination among childrens and adolescents

SECONDARY OUTCOMES:
Proportion of children and adolescents with complete HPV vaccination | 12 months
  Rate of complete HPV vaccination scheme (two doses) among childrens and adolescents
Proportion of teachers with complete HPV vaccination (two doses) | 12 months
  Rate of complete HPV vaccination scheme (two doses) among teachers
Proportion of vaccination refusal among children and adolescents | 12 months
  Rate of HPV vaccination refusal
Proportion of vaccination refusal among teachers | 12 months
  Rate of teacher HPV vaccination refusal

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Henrique A Fonseca, PhD, Study Chair — Academic Research Organization - Hospital Israelita Albert Einstein; Prof. Luiz V Rizzo, PhD, Study Chair — Academic Research Organization - Hospital Israelita Albert Einstein
Locations (79):
- Brazil (79):
  - Cel Filemon Fernandes Teles, Crato, Ceará
  - Dom Vicente de Paula Araujo Matos, Crato, Ceará
  - EEIEF Maria Yara de Brito Gonçalves CAIC, Crato, Ceará
  - EEIF Antonio Antuérpio Gonzaga de Melo, Crato, Ceará
  - EEF José Ferreira Menezes, Juazeiro do Norte, Ceará
  - EEF Raimundo Pessoa, Juazeiro do Norte, Ceará
  - EEF Zila Belem, Juazeiro do Norte, Ceará
  - Emef Mário Da Silva Bem, Juazeiro do Norte, Ceará
  - Emef Professora Maria de Lourdes Lopes de Sousa, Juazeiro do Norte, Ceará
  - EMEIF Maria Do Socorro Cardoso, Juazeiro do Norte, Ceará
  - CED 4 do Guará, Brasília, Federal District
  - CEF 04 Ceilandia, Brasília, Federal District
  - CEF 2 da estrutural, Brasília, Federal District
  - CEF 3 da Estrutural, Brasília, Federal District
  - CEF 4 Guará, Brasília, Federal District
  - CEF Lobo Guará, Brasília, Federal District
  - CEF Santos Dumont, Brasília, Federal District
  - CEF Telebrasília, Brasília, Federal District
  - CEF Vargem Bonita, Brasília, Federal District
  - Cei 02 - Prof João Crisóstomo de Figueiredo, Cuiabá, Mato Grosso
  - Ee Ana Maria Do Couto, Cuiabá, Mato Grosso
  - Ee Mariana Luiza Moreira, Cuiabá, Mato Grosso
  - EE PROFª DIVA HUGUENEY DE SIQUEIRA BASTOS, Cuiabá, Mato Grosso
  - EE PROFº RAFAEL RUEDA, Cuiabá, Mato Grosso
  - Ee Deputado Milton Figueiredo, Várzea Grande, Mato Grosso
  - EE Tancredo de Almeida Neves, Couto de Magalhães de Minas, Minas Gerais
  - EM São Judas Tadeu, Couto de Magalhães de Minas, Minas Gerais
  - EE Arthur Tibães, Diamantina, Minas Gerais
  - EE João Cesar de Oliveira, Diamantina, Minas Gerais
  - EE Professor Gabriel Madacaru, Diamantina, Minas Gerais
  - EE Professor Leopoldo Miranda, Diamantina, Minas Gerais
  - EE Professora Gabriela Neves, Diamantina, Minas Gerais
  - Escola Estadual Professora Isabel Motta, Diamantina, Minas Gerais
  - EE Felício dos Santos, Felício dos Santos, Minas Gerais
  - EM Santo Antônio, Felício dos Santos, Minas Gerais
  - EE Dom João Antônio dos Santo, São Gonçalo do Rio Preto, Minas Gerais
  - EM Zulma Rocha dos Santos, São Gonçalo do Rio Preto, Minas Gerais
  - CE C-M-Ef M Profis Jose Elias da Rocha, Ponta Grossa, Paraná
  - CE Pe-Ef M Pedro Grzelczaki, Ponta Grossa, Paraná
  - CE Prof-Ef M Profis Meneleu A Torres, Ponta Grossa, Paraná
  - CE Prof-Ef M Profis. Joao R V B du Vernay, Ponta Grossa, Paraná
  - EE Profa-Ef Halia T Gruba, Ponta Grossa, Paraná
  - EE-Ef Jesus Divino Operario, Ponta Grossa, Paraná
  - EM Doutor Leopoldo Pinto Rosas, Ponta Grossa, Paraná
  - EM Professora Agenoridas Stadler, Ponta Grossa, Paraná
  - EM Professora Cristiane Levandowski, Ponta Grossa, Paraná
  - EM Professora Zair Santos Nascimento, Ponta Grossa, Paraná
  - EM Professora Zanoni Rogoski, Ponta Grossa, Paraná
  - EM Alfredo Monteiro de Seixas, Augusto Corrêa, Pará
  - EM Andre Alves, Augusto Corrêa, Pará
  - EM Carmem Dilce, Augusto Corrêa, Pará
  - EM Manoel Sady, Augusto Corrêa, Pará
  - EM Maria Benedita Mota, Augusto Corrêa, Pará
  - EM Maria da Conceição Santana, Augusto Corrêa, Pará
  - EM Rosa Athayde, Augusto Corrêa, Pará
  - EM Edom do Nascimento Pinheiro, Tracuateua, Pará
  - EM Elias Ferez Gorayeb, Tracuateua, Pará
  - EM Levina de Oliveira Reis, Tracuateua, Pará
  - EM Valdemar Pinheiro da Silva, Tracuateua, Pará
  - EM Zulmira Guedes, Tracuateua, Pará
  - EE Alceu Amoroso Lima, Natal, Rio Grande do Norte
  - EE Aldo Fernandes, Natal, Rio Grande do Norte
  - EE Djalma Aranha Marinho, Natal, Rio Grande do Norte
  - EE Isabel Gondim, Natal, Rio Grande do Norte
  - EE Reginaldo Ferreira Neto, Natal, Rio Grande do Norte
  - EM Ferreira Itajubá, Natal, Rio Grande do Norte
  - EM José Alves Landim, Natal, Rio Grande do Norte
  - EM José do Patrocínio Pereira Pinto, Natal, Rio Grande do Norte
  - EM Professora Lourdes Godeiro, Natal, Rio Grande do Norte
  - Cem Iii Irmã Maria Teresa Parodi, Boa Vista, Roraima
  - Ee Fagundes Varela, Boa Vista, Roraima
  - Ee Jesus Nazareno de Souza Cruz, Boa Vista, Roraima
  - Em Valdemarina Normando Martins, Boa Vista, Roraima
  - Cem José Aureliano Da Costa, Cantá, Roraima
  - Em Tia Ercília, Cantá, Roraima
  - Cem Maria Mariselma de Oliveira Cruz, Mucajaí, Roraima
  - Ee Vereador Francisco Pereira Lima, Mucajaí, Roraima
  - Em Irmã Leonilde Dal Pós, Mucajaí, Roraima
  - Em Jesus de Nazaré, Mucajaí, Roraima

IPD SHARING:
Plan to Share IPD: No